CLINICAL TRIAL: NCT04985422
Title: Ecological Momentary Intervention for Depressive Symptoms in a Community Sample in Hong Kong: a Randomised Controlled Trial
Brief Title: Ecological Momentary Intervention for Depressive Symptoms in a Community Sample in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Chi-Li Pao Foundation Professor in Psychiatry, Chair Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Flow EMI - Depressive Symptom
Record Dates: First submitted 2021-07-20; First posted 2021-08-02 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Depressive Symptoms
Keywords: Depressive symptoms; Ecological momentary intervention; Rumination; Distress; Stressors; Mental health
MeSH Terms: conditions — Depression; Rumination Syndrome; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Smartphone-based daily ecological momentary intervention (EMI) (Experimental): The experimental group receives 4 weeks of smartphone-based daily EMI. Participants are prompted 6 times a day (with an interval of at least 30 minutes between each digital prompt), on a daily basis over the 4-week period. Within 15 minutes of the digital prompt, participants are to first complete a brief (1-2 minutes) momentary survey ("ecological momentary assessment" [EMA]), and subsequently select 1 out of 5 personalised intervention actions of interest to complete in the moment (time to complete spans from 1 minute to 5 minutes).
  The interventions are brief simple behavioural actions (mostly 1-2 minutes, up to 5 minutes) which could be done in the moment. Simple action tasks include guided breathing, mindful walking, and mindful sound hearing (etc.).
  Participants could also use the platform at any other times to redo intervention actions when preferred. Individualised reports for the EMI completed are provided.
  Interventions: Behavioral: Smartphone-based Daily Ecological Momentary Intervention
- Control group: Smartphone-based weekly-delivered information (Other): The control group receives 4 weeks of smartphone-based weekly-delivered information. The smartphone system (SMS + Qualtrics) as well as the contents of the interventions are identical to those provided to the EMI group. Rather than interventions delivered in the moment on a daily basis over the 4-week period, participants in the control group are provided with a new set of information on a weekly basis over the 4-week period (4 sets in total, 1 new set each week). Participants in the control group are also required to complete a brief 5-minute assessment within 3 days.
  The information includes brief simple behavioural actions (mostly 1-2 minutes, up to 5 minutes) which could be done anytime. Simple action tasks include guided breathing, mindful walking, and mindful sound hearing (etc.).
  Participants could complete any intervention of interest in the information provided at any time throughout the 4-week period.
  Interventions: Behavioral: Smartphone-based Weekly-delivered Information

INTERVENTIONS:
Behavioral: Smartphone-based Daily Ecological Momentary Intervention — Interventions are delivered through smartphones (SMS text message + Qualtrics) at a low cost with high accessibility. Participants are prompted 6 random times a day over the set intervention period (4 weeks) to complete brief EMA and EMI intervention actions) across contexts in daily lives for the reduction of depressive symptoms, as well as rumination distress, and improve functioning.
  Arms: Experimental group: Smartphone-based daily ecological momentary intervention (EMI)
Behavioral: Smartphone-based Weekly-delivered Information — Information with simple actions for reducing depressive symptoms are delivered through smartphones (SMS text message + Qualtrics) at a low cost with high accessibility. Participants are prompted weekly with a new set of information, together with a 5-min assessment. The information includes intervention actions provided in the EMI group.
  Arms: Control group: Smartphone-based weekly-delivered information

SUMMARY:
The key aim of the study is to test the efficacy of a 4-week ecological momentary intervention (EMI), as compared with the regular weekly-based intervention (control group), in reducing (1) symptoms of depression and (2) rumination in community-dwelling individuals. The efficacy of the EMI in reducing distress and improving functioning is also examined.

For both EMI and control groups, the intervention will be delivered through SMS text messages, with a link to a user-friendly and locally-adapted intervention platform designed using Qualtrics (online survey programme).

It is hypothesised that (1) those in the EMI group, as compared to the control group, will show greater reductions in (1) depressive symptoms, (2) rumination level, (3) distress, and in (4) improving functioning. These effects are hypothesised to be observed in individuals with varying levels of symptom severity.

DETAILED DESCRIPTION:
Despite the growth of online-based interventions, there remains a lack of highly adaptive and personalised smartphone-based interventions that can be implemented in the course of everyday life.

The current study examines the effectiveness of a newly-developed smartphone-based ecological momentary intervention (EMI) in reducing symptoms of depression as well as rumination and distress.

Rumination is a common experience in individuals with major depressive disorder (MDD). These psychopathological symptoms occur in a population on a continuous spectrum, which may be especially pronounced after the community has experienced a series of highly stressful and traumatic events. On the high end of the spectrum, manifestations of symptoms may be considered to be clinical disorders, and professional intervention may be indicated. Rumination may affect prognosis and there are suggestions that interventions to reduce and modify rumination can improve outcomes. At the less severe end of the spectrum (i.e., not yet reached the threshold for disorders), rumination may be a risk factor that compromises outcomes and adjustment, one that can cause significant distress and functional impairment. Targeting rumination in both below- and above- threshold populations therefore has important research and clinical implications.

Mental Health Needs in Hong Kong The Hong Kong population has undergone a series of highly stressful events traceable since June 2019, from large-scale social unrest, to the outbreak of Coronavirus disease 2019 (COVID-19) first in January 2020 and a second wave of COVID-19 cases in March 2020. Each of these population-level events is accompanied by other related social, economic, and political consequences, all of which can result in significant psychological distress and mental health burdens especially when added up to individual-level stressors. Local studies have reported heightened depressive symptoms in relation to such population-level events in addition to personal stressful events. The rates observed are considerably higher than the average global prevalence, which marks it as particularly concerning when help-seeking is severely minimal in the general local population. It is anticipated that these rates will continue rising and would manifest with symptoms of other conditions (such as anxiety, as is already seen in China during COVID-19). Unsurprisingly, the widespread pandemic has already led researchers in many other countries to call for enhanced and novel psychological interventions.

A local online self-help initiative has recently been launched by the Department of Psychiatry of the University of Hong Kong, offered to individuals via different channels (including various social media platforms, non-governmental organisations, social and personal connections) in the form of an anonymous mental health recognition and support tool. The key aims of the tool are to provide users with a space to reflect on the ongoing events in their lives and their feelings, provide them with an individualised understanding of their current mental health conditions (MDD symptoms) and the potential contributing factors, as well as offer individualised suggestions for self-help and professional help when necessary. A high level of MDD as well as significant levels of rumination in response to the community stressors have been reported, particularly in young people. Of importance, rumination about such large-scale external events ("event-based rumination") was seen to be highly associated with MDD symptoms.

Rumination and its Consequences In the presence of significant external stressors, an excessive level of symptoms, together with rumination about the stressors or their psychological responses characterise a state described as adjustment disorder (AjD) in the International Classification of Diseases, 11th Revision (ICD-11). The presence of AjD carries an increased level of risk for transition into other clinical disorders, such as MDD. The role of rumination as a mechanism that predisposes individuals towards the development of major depressive episodes has been well studied. Researchers have shown that particular types of rumination, such as brooding (i.e., passive and judgmental comparison of current situation and an unachieved alternative outcome), are specifically responsible for the development of depression. The presence of this rumination type for people with MDD also predicted poorer outcomes. Because of its importance, interventional strategies (such as cognitive-behavioural therapy, CBT) targeting rumination have been developed and have been shown to be effective in improving mental health outcomes. Rumination-focused CBT generally involves increasing one's ability to become aware of their own (brooding) ruminations and supporting them to eventually replace them with alternative thinking habits).

Ecological Momentary Assessment and Intervention Recent years have seen the growth of a new avenue for mental health that appears highly suitable for the Hong Kong population, namely ecological momentary assessment (EMA) and ecological momentary intervention (EMI). These mobile health (mHealth) approaches offered new opportunities for mental health research, management, detection, and intervention via smartphones. In EMA, individuals can self-initiate assessments when an emotion or specific event is experienced (event-sampling), or are prompted several times a day to complete brief assessments over a number of days (time-sampling). While EMIs have been used to augment usual treatments, EMIs have also been coupled with EMA to deliver interventions based on symptoms reported in the moment. The essence of these two approaches is their abilities to be implemented in real-time and in everyday life contexts, be designed flexibly according to specific objectives, and be adapted to individual needs. Capturing prospective information on interactions between micro-level experiences and real-world contexts, as well as providing in-the-moment interventions, EMA and EMI impart benefits that cannot be achieved in traditional in-person treatments.

Importantly, increasing evidence from randomised controlled trials (RCTs) has shown EMI to be an efficacious and effective means to augment interventions in different disorders, including depression, anxiety, bipolar disorders, psychosis. Furthermore, although EMA in addition to treatment-as-usual (TAU) has shown to be more effective than TAU alone in reducing depressive symptoms in patients with MDD, the positive impact of EMI was shown to be more long-lasting in the EMI+TAU group compared with EMI+TAU, with the effects lasting for up to 3 months for EMA+TAU, and up to 6 months for EMI+TAU.

The Current Study EMI appears to be a promising approach to support individuals with distress in the Hong Kong population in reducing symptoms and ruminative thoughts. This is also possibly the only means to reach those less motivated to seek help due to stigma, as well as potential worries over in-person contacts especially after the COVID-19 outbreak.

The key aim of the study is to test the efficacy of a 4-week ecological momentary intervention (EMI), as compared with the regular weekly-based intervention (control group), in reducing (1) symptoms of depression and (2) rumination in community-dwelling individuals. The efficacy of the EMI in reducing distress and improving functioning is also examined.

It is hypothesised that (1) those in the EMI group, as compared to the control group, will show greater reductions in (1) depressive symptoms, (2) rumination level, (3) distress, and in (4) improving functioning. These effects are hypothesised to be observed in individuals with varying levels of symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of depression indicated by DASS-D score of 10 or above
* Aged 15 to 64 years (parental or guardian consent is required for those below 18 years)
* Possess a smartphone with access to the Internet

Exclusion Criteria:

* Significant developmental disorder, psychotic disorder, substance abuse or organic brain disorder
* Active suicidal risk
* Receiving active structured intervention or anticipating to receive such treatment (e.g., biweekly psychotherapy sessions, receiving pharmacotherapy)

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 262 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms, as assessed using the Depression subscale of the Depression, Anxiety and Stress Scales (DASS-D) | Immediately after intervention (post 4-week intervention) and up to 3 months
  The DASS-D is a 7-item measure rated on a 4-point Likert scale. Scores range from 0 to 42, where a higher score represents a higher level of depressive symptoms. The DASS-D has been validated in Hong Kong (epidemiological and clinical samples) as well as in both young people and adults.

SECONDARY OUTCOMES:
Change in rumination level, as assessed using the 10-item ruminative response scale (RRS-10) | Immediately after intervention (post 4-week intervention) and up to 3 months
  The RRS-10 is a 10-item measure rated on a 4-point Likert scale. Scores range from 10 to 40, where a higher score represents a higher level of ruminative experience.
Change in psychological distress, as assessed using the Kessler Psychological Distress Scale (K6) | Immediately after intervention (post 4-week intervention) and up to 3 months
  The K6 is a 6-item measure rated on a 5-point Likert scale. Scores range from 0 to 24, where a higher score represents a higher level of distress symptoms.
Change in level of functioning, as reflected by presenteeism and absenteeism due to distress | Immediately after intervention (post 4-week intervention) and up to 3 months
  Presenteeism is assessed using an item that asks the number of days during the past four weeks the participant has to cut down on work, study, or manage day-to-day activities due to distress. Absenteeism is assessed using an item that asks the number of days during the past four weeks the participant has been totally unable to work, study, or manage day-to-day activities due to distress.

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Chen, MA, Principal Investigator — The University of Hong Kong; Stephanie MY Wong, BSocSc, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Lam LC, Chan WC, Wong CS, Chen EY, Ng RM, Lee EH, Chang WC, Hung SF, Cheung EF, Sham PC, Chiu HF, Lam M, Chiang TP, van Os J, Lau JT, Lewis G, Bebbington P; Hong Kong Mental Morbidity Survey Team. The Hong Kong mental morbidity survey: background and study design. East Asian Arch Psychiatry. 2014 Mar;24(1):30-6. PMID 24676485
- [Background] Echiverri AM, Jaeger JJ, Chen JA, Moore SA, Zoellner LA. "Dwelling in the Past": The Role of Rumination in the Treatment of Posttraumatic Stress Disorder. Cogn Behav Pract. 2011 Aug;18(3):338-349. doi: 10.1016/j.cbpra.2010.05.008. PMID 22190846
- [Background] Nolen-Hoeksema S, Wisco BE, Lyubomirsky S. Rethinking Rumination. Perspect Psychol Sci. 2008 Sep;3(5):400-24. doi: 10.1111/j.1745-6924.2008.00088.x. PMID 26158958
- [Background] Watkins ER. Constructive and unconstructive repetitive thought. Psychol Bull. 2008 Mar;134(2):163-206. doi: 10.1037/0033-2909.134.2.163. PMID 18298268
- [Background] Ni MY, Yao XI, Leung KSM, Yau C, Leung CMC, Lun P, Flores FP, Chang WC, Cowling BJ, Leung GM. Depression and post-traumatic stress during major social unrest in Hong Kong: a 10-year prospective cohort study. Lancet. 2020 Jan 25;395(10220):273-284. doi: 10.1016/S0140-6736(19)33160-5. Epub 2020 Jan 9. PMID 31928765
- [Background] Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, Ho RC. Immediate Psychological Responses and Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19) Epidemic among the General Population in China. Int J Environ Res Public Health. 2020 Mar 6;17(5):1729. doi: 10.3390/ijerph17051729. PMID 32155789
- [Background] Wind TR, Rijkeboer M, Andersson G, Riper H. The COVID-19 pandemic: The 'black swan' for mental health care and a turning point for e-health. Internet Interv. 2020 Apr;20:100317. doi: 10.1016/j.invent.2020.100317. Epub 2020 Mar 19. No abstract available. PMID 32289019
- [Background] Wong SMY, Hui CLM, Wong CSM, Suen YN, Chan SKW, Lee EHM, Chang WC, Wong GHY, Chen EYH. Induced ideas of reference during social unrest and pandemic in Hong Kong. Schizophr Res. 2021 Mar;229:46-52. doi: 10.1016/j.schres.2021.01.027. Epub 2021 Feb 19. PMID 33618286
- [Background] Wong SM, Hui CL, Wong CS, Suen YN, Chan SK, Lee EH, Chang WC, Chen EY. Prospective prediction of PTSD and depressive symptoms during social unrest and COVID-19 using a brief online tool. Psychiatry Res. 2021 Apr;298:113773. doi: 10.1016/j.psychres.2021.113773. Epub 2021 Jan 29. PMID 33545423
- [Background] Wong SMY, Hui CLM, Wong CSM, Suen YN, Chan SKW, Lee EHM, Chang WC, Chen EYH. Mental Health Risks after Repeated Exposure to Multiple Stressful Events during Ongoing Social Unrest and Pandemic in Hong Kong: The Role of Rumination: Risques pour la sante mentale apres une exposition repetee a de multiples evenements stressants d'agitation sociale durable et de pandemie a Hong Kong: le role de la rumination. Can J Psychiatry. 2021 Jun;66(6):577-585. doi: 10.1177/0706743720979920. Epub 2020 Dec 15. PMID 33317325
- [Background] Myin-Germeys I, Kasanova Z, Vaessen T, Vachon H, Kirtley O, Viechtbauer W, Reininghaus U. Experience sampling methodology in mental health research: new insights and technical developments. World Psychiatry. 2018 Jun;17(2):123-132. doi: 10.1002/wps.20513. PMID 29856567
- [Background] Kramer I, Simons CJ, Hartmann JA, Menne-Lothmann C, Viechtbauer W, Peeters F, Schruers K, van Bemmel AL, Myin-Germeys I, Delespaul P, van Os J, Wichers M. A therapeutic application of the experience sampling method in the treatment of depression: a randomized controlled trial. World Psychiatry. 2014 Feb;13(1):68-77. doi: 10.1002/wps.20090. PMID 24497255